CLINICAL TRIAL: NCT00775229
Title: A Double-blind, Placebo-controlled Study of Naltrexone in Trichotillomania
Brief Title: Naltrexone in the Treatment of Trichotillomania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0806M36061
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Results first posted 2014-03-17 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Trichotillomania
Keywords: hair pulling
MeSH Terms: conditions — Trichotillomania | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Naltrexone
  Interventions: Drug: Naltrexone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — pill, by mouth, 50mg-150mg/day for the duration of the study
  Other Names: ReVia
  Arms: 1
Drug: Placebo — pill, by mouth, daily
  Other Names: also known as a 'sugar pill'
  Arms: 2

SUMMARY:
This is an 8-week, double-blind study of Natrexone in the treatment of trichotillomania

DETAILED DESCRIPTION:
The goal of the proposed study is to evaluate the efficacy of Naltrexone in trichotillomania. Forty subjects with DSM-IV trichotillomania will receive 8 weeks of double-blind Naltrexone or placebo. The hypothesis to be tested is that Naltrexone will be effective and well tolerated in patients with trichotillomania compared to placebo. The proposed study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

ELIGIBILITY:
Inclusion Criteria:

1. men and women age 18-75;
2. current DSM-IV trichotillomania;
3. hair-pulling primarily due to urges/cravings; and 4) pulling is reported as pleasurable the majority of time.

Exclusion Criteria:

1. unstable medical illness or clinically significant abnormalities on pre-study laboratory tests or physical examination;
2. history of seizures;
3. myocardial infarction within 6 months;
4. current pregnancy or lactation, or inadequate contraception in women of childbearing potential;
5. clinically significant suicidality;
6. current or recent (past 3 months) DSM-IV substance abuse or dependence;
7. illegal substance within 2 weeks of study initiation;
8. initiation of psychotherapy or behavior therapy from a mental health professional for the treatment of trichotillomania within 3 months prior to study baseline;
9. initiation of a psychotropic medication within 2 months prior to study inclusion;
10. previous treatment with naltrexone; and
11. treatment with investigational medication or depot neuroleptics within 3 months, with fluoxetine within 6 weeks, or with other psychotropics within 2 weeks prior to study baseline;
12. lifetime history of DSM-IV bipolar disorder type I, dementia, or schizophrenia or any other DSM-IV psychotic disorder;
13. current use of opiates.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-08; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Hoffman J, Williams T, Rothbart R, Ipser JC, Fineberg N, Chamberlain SR, Stein DJ. Pharmacotherapy for trichotillomania. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD007662. doi: 10.1002/14651858.CD007662.pub3. PMID 34582562
- [Derived] Odlaug BL, Chamberlain SR, Harvanko AM, Grant JE. Age at onset in trichotillomania:clinical variables and neurocognitive performance. Prim Care Companion CNS Disord. 2012;14(4):PCC.12m01343. doi: 10.4088/PCC.12m01343. Epub 2012 Jul 19. PMID 23251869

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men and women aged 18 to 75 years with a primary Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis of TTM were recruited through newspaper advertisements and referrals.
Pre-assignment Details: Exclusion: unstable medical illness, current pregnancy or inadequate contraception, thoughts of suicide,history of bipolar disorder,dementia, or psychotic disorder,past 12 months SUD, previous treatment with naltrexone, initiation of behavior therapy within the last 6 months, initiation of a psychotropic medication within the last 3months, opiates.
Groups:
- Naltrexone: Naltrexone
  Naltrexone : pill, by mouth, 50mg-150mg/day for the duration of the study
- Placebo: Placebo
  Placebo : pill, by mouth, daily
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 25 | 26
Completed | 20 | 24
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 26 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (9.4) | 34.0 (10.1) | 32.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: National Institute of Mental Health Trichotillomania Symptom Severity Scale
Description: Ranges from 0-20 with 20 being the most severe. The lower the total score, the lower the severity level. This scale is given and measured once every 2 weeks for a total of 8 weeks. The final total score is reported here.
Time Frame: This is the final score, measured at week 8 (final visit).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 25 | 26
units on a scale | 7.94 (4.835) | 8.73 (5.481)

2. Secondary Outcome: Massachusetts General Hospital Hairpulling Scale
Description: Ranges from 0-28 with 28 being the most severe. The lower the total score, the lower the severity level. This scale is given and measured once every 2 weeks for a total of 8 weeks. The final total score is reported here.
Time Frame: This is the final score, measured at week 8 (final visit).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 25 | 26
units on a scale | 12.21 (6.203) | 13.35 (4.749)

3. Secondary Outcome: Liver Function Tests
Description: Participants were administered a general test of liver functioning to asses safety over the course of the study. Data represent the percentage of participates with Liver Function Test values falling outside of the range considered safe/typical for liver functioning at any of the assessed time points. It was performed at baseline and at each visit where dosage of the medication is >50mg/day (week 2-week 8).
Time Frame: Week 8 (last visit)
Measure: Number; unit: percentage of individuals with LFT chang
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 25 | 26
percentage of individuals with LFT chang | 0 | 0

ADVERSE EVENTS:
Arm/Group | Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 3/25 | 1/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=25) | Placebo (N=26)
Sedation (Psychiatric disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No